CLINICAL TRIAL: NCT06315075
Title: Dialectical Behavior Therapy for Adolescents With Self-harm and Suicidal Behavior- an Open
Brief Title: Dialectical Behavior Therapy for Adolescents With Self-harm and Suicidal Behavior- an Open Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 657876
Record Dates: First submitted 2024-02-27; First posted 2024-03-18 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Self-harm; Suicidal Ideation; Suicide and Self-harm
Keywords: Suicide and Self-harm; Adolescents; Dialectical behavior therapy for adolescents; Routine clinical practice; Effectiveness study
MeSH Terms: conditions — Self-Injurious Behavior; Suicidal Ideation; Suicide | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Single group, uncontrolled, pre-post-one year follow-up study
Masking Description: An independent evaluator will assess participants at post treatment and one year follow-up. Due to the single group design, the assessor will be aware that participants have received the intervention, but will not be involved in recruitment and treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBT-A (Experimental): Single group uncontrolled study. All participants will receive DBT-A
  Interventions: Behavioral: Dialectical behavior therapy for adolescents (DBT-A)

INTERVENTIONS:
Behavioral: Dialectical behavior therapy for adolescents (DBT-A) — A 20-week DBT-A with a weekly individual session (45 minutes), a weekly session of multifamily skills training groups with a caregiver (120 minutes), and telephone consultation with individual therapists outside therapy sessions as needed. The treatment consists of four components and is delivered according to the manual except for the phone coaching that PBU offers workdays until 8 pm.
  Other Names: DBT-A

SUMMARY:
The goal of this pre-post-follow-up study is to examine how well the treatment Dialectical behavior therapy for adolescents (DBT-A) with a duration of 20 weeks for adolescents with self-harm and suicidal behavior works in routine clinical practice. The main questions it aims to answer are:

* to investigate how well DBT-A works after treatment and at 3-month follow-up, measured by episodes of self-harm, suicide attempts, depressive symptoms and quality of life, drop-out from treatment and number of possible participants who decline DBT-A.
* to investigate how well DBT-A works at 12 months follow-up
* to investigate whether pre-treatment factors can predict who will benefit from treatment

DETAILED DESCRIPTION:
Self-harm and suicidal ideation are prevalent among adolescents and associated with major mental health problems and adverse life events. Dialectical behavior therapy for adolescents (DBT-A) is an empirically supported treatment for self-harm and suicidal ideation in adolescents. However, knowledge is scarce on the effectiveness, long-term outcomes, acceptability, and dropout of DBT-A when implemented and delivered as part of routine clinical practice in the Norwegian national health care system. The main aim of this study is to examine the outcomes from DBT-A in terms of self-harm episodes, suicide attempts, and emergency hospital admission, in addition to acceptability and dropout, when DBT-A is delivered at the Department of Child and adolescent psychiatry (PBU), Haukeland University Hospital (HUS). The study is an uncontrolled pre-post study with one-year follow-up and includes three aims: to evaluate outcomes of DBT-A up to three months post-treatment, at one-year follow-up, and to describe predictors of outcome for adolescents receiving DBT-A.

ELIGIBILITY:
Inclusion Criteria:

* Age 13-18 years
* Ongoing or a history of self-harm the last six months; current suicidal behavior (suicidal thoughts or at least one suicide attempt within the previous six months); at least three criteria of Diagnostic and Statistical Manual -5 (DSM-5) Borderline personality disorder (BPD), or the self-destruction criterion of DSM-5 BPD in addition to minimum two subthreshold criteria as assessed by the Structured Clinical Interview for DSM-5 Personality Disorders (SCID-5-PD) (First et al., 2016)
* Fluency in Norwegian
* One parent/trusted adult that can participate together with the adolescent.

Exclusion Criteria:

* Intellectual disability
* Significant learning or language impairments
* Autism spectrum disorder
* Anorexia Nervosa
* Any psychotic disorder
* Substance abuse disorder. These patients will be offered treatment as usual at their local outpatient clinic.

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Lifetime Parasuicide Count Interview | pre, after 20 weeks DBT-A ("post"), at 3 and 12 months follow-up
  Number of self-harm episodes in the last four weeks categorized by intention and self-harm method, number of suicide attempts, and number of emergency department visits caused by suicidal behavior.
Number of participants in need of emergency department visits caused by suicidal behavior | pre, after 20 weeks DBT-A ("post"), at 3 and 12 months follow-up
  Medical record data extraction

SECONDARY OUTCOMES:
Depressive symptom score measured by Short Mood and Feelings questionnaire (SMFQ) | pre, after 20 weeks DBT-A ("post"), 3 and 12 months follow-up
  Depressive symptoms. SMFQ includes 13 items, measured on a 0-2 Likert scale, with higher scores indicating a higher level of depressive symptoms.
Health related quality of life measured by SCREENing for and Promotion of Health Related Quality of Life in Children an Adolescents (Kidscreen 10) | pre, after 20 weeks DBT-A ("post"), 3 and 12 months follow-up
  Kidscreen includes 10 items measured on a 5 point Likert scale and gives a global measure from 0-100 of health-related quality of life in addition to the individual aspects. Higher scores reflects higher health related quality of life.
Barriers to Treatment Participation Scale (BTPS) score | pre, at dropout at any time between session 1 and end of treatment at session 20.
  The BTPS questionnaire evaluate reasons for treatment discontinuation, and treatment participation barriers.
Perceived benefit of skills training in DBT-A measured by a study specific questionnaire. | At dropout at any time between session 1 and end of treatment at session 20, or for completers after 20 weeks DBT-A ("post"),
  Perceived benefit of skills training in DBT-A is a study-specific patient- and parent reported evaluation measure of perceived benefits of DBT-A components rated on a 0-5 Likert scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gro Janne H. Wergeland, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (1):
- Dept. of child and adolescent psychiatry, Haukeland University Hospital, Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No